CLINICAL TRIAL: NCT04223596
Title: Clinical Utility of Liquid Biopsy as a Tool to Assess the Evolution of Brigatinib Treated Patients With Non-small Cell Lung Cancer With EML4-ALK Translocation: an Exploratory Study
Brief Title: Clinical Utility of Liquid Biopsy in Brigatinib ALK+ Patients
Acronym: CUBIK
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación GECP (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GECP 19/01_CUBIK; 2019-002369-36 (EudraCT Number)
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Lung Cancer; NSCLC; NSCLC Stage IIIB; NSCLC Stage IV
Keywords: Lung cancer; ALK +; locally advanced; metastasic SCLC; brigatinib; non small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — brigatinib

STUDY DESIGN:
Intervention Model Description: Open-label, non-randomised, phase II, exploratory, multi-country and multi-centre clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Brigatinib Arm (Experimental): Brigatinib 90 mg for the first 7 days and then 180 mg daily thereafter for QW4 cycles of duration (28 days +- 3 days)
  Interventions: Drug: Brigatinib

INTERVENTIONS:
Drug: Brigatinib — Brigatinib 90 mg for the first 7 days (D1-7 at cycle 1) and then 180 mg daily thereafter for QW4 cycles of duration (28 days+-3 days)
  Other Names: AP26113

SUMMARY:
This is an open-label, non-randomised, phase II, exploratory, multi-country and multi-centre clinical trial. Chemotherapy-naïve patients with EML4-ALK rearrangement and with locally advanced or metastatic non-small cell lung cancer patients will be selected.

Patients enrolled in the study will receive brigatinib 90mg for the first 7 days (D 1-7 at cycle 1) and then 180mg daily thereafter for QW4 cycles of duration (28 days ±3days).

Brigatinib will be administered until progression disease, unacceptable toxicity, patient or physician decision to discontinue or death.

Brigatinib may continue beyond disease progression per RECIST v1.1 until loss of clinical benefit, unacceptable toxicity, patient or physician decision to discontinue, or death as per SmPC recommendations.

Patient accrual is expected to be completed within 1.5 years excluding a run-in-period of 4-6 months. Treatment and follow-up are expected to extend the study duration to a total of 5 years. Patients will be followed for 1 year after the end of treatment independently of the cause of end of treatment. The study will end once survival follow-up has concluded.

The trial will end with the preparation of the final report, scheduled for 5.5 years after the inclusion of the first patient approximately.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥ 18 years old
2. ECOG performance status of 0-2
3. Histologically or cytologically confirmed, Stage IIIB or IV NSCLC according to 8th version of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology, that is ALK+
4. Patients who have documented locally ALK rearrangement by one of the following methods:

   1. a positive result from the Vysis® ALK Break-Apart fluorescence in situ hybridization (FISH) Probe Kit; or
   2. IHC with VENTANA ALK (D5F3) CDx assay
5. No prior treatment for Stage IIIB or IV non-squamous NSCLC.
6. Having a life expectancy ≥ 3 months
7. Patients who have received prior neo-adjuvant, adjuvant chemotherapy, radiotherapy, or chemo-radiotherapy with curative intent for non-metastatic disease must have experienced a treatment-free interval of at least 6 months from enrollment since the last chemotherapy, radiotherapy, or chemo-radiotherapy.
8. Untreated or treated CNS metastases allowed, as long as asymptomatic and neurologically stable
9. Patients with at least 1 measurable lesion, as defined by RECIST v1.1. Previously irradiated lesions can only be considered as measurable if disease progression has been unequivocally documented at that site since radiation and the previously irradiated lesion is not the only site of disease.
10. Normal QT interval (QT) on screening ECG evaluation, defined as QT interval corrected (Fridericia) (QTcF) of ≤ 450 milliseconds (msec) in males of ≤ 470 msec in females
11. Adequate hematologic and organ function defined by the following laboratory results obtained within 14 days prior to enrollment:

    * (ANC) Neutrophils ≥ 1500 cells/μL without granulocyte colony-stimulating factor support.
    * Lymphocyte count ≥ 500/μL.
    * Platelet count ≥ 75,000/μL without transfusion.
    * Haemoglobin ≥ 10.0 g/dL.
    * INR or aPTT ≤ 1.5 × upper limit of normal (ULN). This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose.
    * AST, ALT, and alkaline phosphatase ≤ 2.5 × ULN, with the following exceptions:

    Patients with documented liver metastases: AST and/or ALT ≤ 5 × ULN. Patients with documented liver or bone metastases: alkaline phosphatase ≤ 5 × ULN.
    * Serum bilirubin ≤ 1.5 × ULN. Patients with known Gilbert disease who have serum bilirubin level < 3 × ULN may be enrolled.
    * Serum creatinine ≤ 1.5 × ULN
    * Serum lipase and amylase ≤ 1.5 × ULN
12. All patients are notified of the investigational nature of this study and signed a written informed consent in accordance with institutional and national guidelines, including the Declaration of Helsinki prior to any trial-related intervention.
13. Willingness and ability to comply with scheduled visits and study procedures
14. For female patients of childbearing potential, a negative pregnancy test must have been documented prior to enrollment (within 14 days prior to enrollment)
15. For female patients of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception that results in a low failure rate (< 1% per year) when used consistently and correctly, and to continue its use for 4 months after the last dose of brigatinib. No hormonal methods and preferably barrier method always containing a spermicide, intrauterine device (IUD): intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner (on the understanding that this is the only one partner during the whole study duration), and sexual abstinence.
16. For male patients with female partners of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception that results in a low failure rate [< 1% per year] when used consistently and correctly, and to continue its use for 4 months after the last dose of brigatinib. Male patients should not donate sperm during this study and for at least 4 months after the last dose of brigatinib.
17. Women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile must have a negative serum pregnancy test result within 14 days prior to enrollment.

Exclusion Criteria:

1. Patients with a known sensitizing mutation in the epidermal growth factor receptor (EGFR) gene.
2. Patients with a known STK-1 Ligand alteration.
3. Patients with a known MDM2 amplification.
4. Patients with a known ROS1 translocations.
5. Patients that received any prior TKI, including ALK-targeted TKIs or any systemic anticancer therapy for locally advanced or metastasic disease
6. Patients that have received chemotherapy or radiation within 14 days of first dose of study drug, except stereotactic radiosurgery (SRS) or stereotactic body radiation therapy (SBRT)
7. Symptomatic CNS metastases (parenchymal or leptomeningeal) that are neurologically unstable or required an increasing dose of corticosteroids within 7 days prior to first dose of study drug
8. Have current spinal cord compression (symptomatic or asymptomatic and detected by radiographic imaging). Patients with leptomeningeal disease and without cord compression is allowed.
9. Malignancies other than NSCLC within 3 years prior to enrollment (except for adequately treated non-melanoma skin cancer, carcinoma in situ of the cervix, localized prostate cancer treated surgically with curative intent, which were allowed within 3 years)
10. Women who are pregnant, lactating, or intending to become pregnant during the study.
11. Patients that received monoclonal antibodies or had major surgery within 30 days of the first dose of brigatinib (Day 1, Cycle1) or anticipation of need for a major surgical procedure during the course of the study.
12. History of idiopathic pulmonary fibrosis, pulmonary interstitial disease, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
13. Have uncontrolled hypertension. Patients with hypertension should be under treatment on study entry to control blood pressure.
14. Positive test for HIV. All patients will be tested for HIV prior to inclusion into the study; patients who test positive for HIV will be excluded from the clinical study.
15. Patients with active hepatitis B (chronic or acute; defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C.

    * Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBcAb] and absence of HBsAg) are eligible only if they are negative for HBV DNA.
    * Patients positive for hepatitis C virus (HCV) antibody are eligible only if PCR is negative for HCV RNA.
16. Active tuberculosis.
17. Severe infections within 2 weeks prior to be included in the study, including but not limited to hospitalization for complications of infection, bacteraemia, or severe pneumonia.
18. Have significant, uncontrolled or active cardiovascular disease specifically including but not restricted to:

    * such as New York Heart Association cardiac disease (Class II or greater),
    * myocardial infarction (MI) within 6 months prior to the first dose of study drug
    * unstable angina within 6 months prior to the first dose of study drug
    * congestive heart failure (CHF) within 6 months of the first dose of study drug
    * history of clinically significant atrial arrhythmia (including clinically significant bradyarrhythmia), as determined by the treating physician
    * any history of ventricular arrhythmia
    * cerebrovascular accident or transient ischemic attack within 6 months prior to the first dose of study drug NOTE: Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate.
19. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the patient at high risk from treatment complications.
20. Patients with illnesses or conditions that interfere with their capacity to understand follow and/or comply with study procedures.
21. History of or active significant GI bleeding or coagulopathy (in the absence of therapeutic anticoagulation) within 3 months of the first dose of brigatinib
22. History of blood transfusion within 3 months of blood draw for translational research
23. Malabsorption syndrome or other GI illness that could affect oral absorption of the study drug
24. Evidence of abdominal free air not explained by paracentesis or recent surgical procedure.
25. Serious, non-healing wound, active ulcer, or untreated bone fracture
26. Known or suspected hypersensitivity to brigatinib or its excipients
27. Evidence of any other disorder or significant laboratory finding that makes the patient undesirable to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | From date of randomization until the date of first documented progression or date of death, whichever came first, assessed up to 60 months
  To evaluate the Overall response rate of brigatinib as measured by investigator. It will be assessed per RECIST v1.1 criteria. ORR is defined as the proportion of patients who have a partial or complete response to therapy; it does not include stable disease and is a direct measure of drug tumoricidal activity.

SECONDARY OUTCOMES:
Duration of response (DOR) | From date of documentation of tumor response until date of first documented progression, assessed up to 60 months.
  To evaluate the efficacy of brigatinib as measured by investigator. Assessed as duration of response (DOR) according to RECIST v1.1
Intracranial overall response rate (ORR) | From date of documentation of tumor response until date of first documented progression, assessed up to 60 months.
  To evaluate the intracranial ORR defined as the proportion of patients with reduction in intracranial tumor
Progression free survival (PFS) rate | 1 year and 2 years of treatment with Brigatinib
  To evaluate PFS rate until first progression documented during the treatment with brigatinib by RECIST v1.1
Overall Survival (OS) rate | 1 year and 2 years of treatment with Brigatinib
  To evaluate the OS defined as the lenght of time from either the date of diagnosis or the start of the treatment that patients diagnosed with the disease are still alive.
Safety and tolerability: NCI CTCAE v4.0 criteria | From the subject's written consent to participate in the study through 30 days after the final administration of the drug.
  Occurrence and severity of adverse events, with severity determined by NCI CTCAE v4.0 criteria.
Time on treatment (TTR) | From date of the start of treatment until first objective tumour response observed (partial or complete according RECIST v1.1), assessed up to 60 months.
  To evaluate the efficacy of brigatinib as measured by investigator according to RECIST v1.1. TTR is defined as the time from the start of treatment to the first objective tumour response observed for patients who achieved Complete Response or Partial Response (according RECIST v.1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Provencio, MD, Principal Investigator — Fundación GECP President
Locations (15):
- Spain (15):
  - Complejo Hospitalario de A Coruña, A Coruña, A Coruña
  - Hospital General de Alicante, Alicante, Alicante
  - Hospital Regional Universitario de Málaga, Málaga, Andalusia
  - Hospital Son Espases, Palma de Mallorca, Balearic Islands
  - ICO Badalona, Badalona, Barcelona
  - ICO Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Universitario Insular de Gran canaria, Las Palmas de Gran Canaria, Gran Canaria
  - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Puerta de Hierro, Madrid, Madrid
  - Hospital Clínico de Salamanca, Salamanca, Salamanca
  - Hospital Universitari i Politécnic La Fe, Valencia, Valencia
  - Hospital General de Valencia, Valencia, Valencia
  - Hospital Universitario de Cruces, Barakaldo, Vizcaya
  - Hospital Vall Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: fundación GECP page — http://www.gecp.org